CLINICAL TRIAL: NCT06735846
Title: Clinical Investigation to Evaluate the Safety and Performance of Demax Guide Wire
Brief Title: Single Arm, Prospective, Open-label, Multi-center Clinical Investigation for the Demax Guide Wire
Acronym: SPOMCIDGW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DemaxGroup (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DMK/QS-QP32-QD03.15-TJ
Record Dates: First submitted 2024-11-10; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Vascular Diseases; Coronary Artery Disease
MeSH Terms: conditions — Peripheral Vascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Demax Guide Wire (Experimental): The objectives of this study are to confirm the safety and performance of the Guide Wire when used in patients with peripheral vasculature or coronary vasculature disease.
  Interventions: Device: Guide wire

INTERVENTIONS:
Device: Guide wire — Insert the distal end of the guide wire into the introducer sheath and enter the blood vessel through the introducer sheath;5.Insert the catheter directly into the blood vessel through the guide wire, and when the catheter reaches the target position, exit the guide wire.

SUMMARY:
The objectives of this study are to confirm the safety and performance of the Guide Wire when used in patients with peripheral vascular or coronary vascular disease for diagnostic or treatment procedures and will be the pivotal trial for this device. This study intends to evaluate the Guide Wire in its ability to successfully deploy an intended diagnostic or therapeutic catheter according to the IFU without any device related deficiencies, time to reach a specified position, and total number of insertion attempts to reach a primary performance endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 18 years old or older
2. Written consent to participate in the study
3. All subjects must be candidates to undergo percutaneous peripheral or coronary diagnostic or interventional procedures where use of a Guide Wire is indicated.
4. Eligible for catheter-based diagnostic or treatment procedure. A representative list of diseases and catheter-based treatments includes:

   Suspicion of obstructive coronary artery disease manifest as myocardial infarction, angina pectoris, angina-equivalent, ischemic dysrhythmia, or evidence of ischemia or viability on non-invasive cardiovascular testing Suspicion of peripheral vascular obstructive disease undergoing elective or urgent diagnostic and/or percutaneous therapeutic procedures.
5. Palpable pulse of the proximal and distal radial artery on one or both arms
6. Subjects must be suitable for a transfemoral vascular access
7. Subjects undergoing elective or urgent percutaneous treatment of symptomatic arterial occlusive disease and intermittent claudication or CLI of the SFA and/or popliteal arteries.
8. Subjects with suspected narrowed or blocked arteries in the heart.

Exclusion Criteria:

1. Inability to provide consent
2. Pregnant or lactating women
3. Subjects actively participating in another drug or device investigational study and have not yet completed the primary endpoint follow-up period.
4. Subjects with bilateral hand or arm misalignment / paresis that makes a radial access impossible
5. Subject has a known allergy to the Guide Wire materials
6. Subjects with emergent procedures acute ischemia, aneurysmal disease, common femoral or profunda interventions, or hybrid procedures were excluded.
7. Subjects with severe infections
8. Subjects with severe heart failure
9. Subjects with severe physical weakness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | up to 15 ± 2 days after the procedure.
  Freedom from SADEs during the procedure and up to 15 ± 2 days after the procedure.
Primary Performance Endpoint | Catheter according to the IFU, insertion attempt to reach deployment(up to< 24 hours)
  Successful introduction of Guide Wire and deployment of the intended diagnostic or therapeutic catheter according to the IFU, without any device related deficiencies per insertion attempt

SECONDARY OUTCOMES:
Rate of Guide Wire deficiencies; | 15 ± 2 days after the procedure
  Any inadequacy in the identity, quality, durability, reliability, safety or performance of an investigational device, including malfunction, use errors or inadequacy in information supplied by the manufacturer. In regard to guide wire deficiencies, once captured, we will compare the rate of guide wire deficiencies to the rates of occurrence outlined within the risk management file to see if they match. If the Guidewire deficiencies are over what is found in the risk management file this could lead to a change in risk mitigation.
Rate of complications: | 15 ± 2 days after the procedure
  Air embolism, Arteriovenous fistula, Infection, Ischemia, Death, Myocardial infarction, Perforation of the vessel wall, Hematoma at the puncture site, Stroke or system embolization, Thrombus formation, Vascular dissection, Vasospasm
Expected number of insertion attempts for a single Guide Wire to reach primary performance endpoint | Catheter according to the IFU, insertion attempt to reach deployment(up to< 24 hours)
  It is designed to capture the total number of insertion attempts, it can only be qualitative due each procedure being different. Variables for each procedure include (but not limited) the following: Clinical condition of patient, product type used, point of entry site, skill of user.
Expected time to reach the specified position with the Guide Wire | Catheter according to the IFU, insertion attempt to reach deployment(up to< 24 hours)
  It is designed to consider the subjective nature of time taken during the procedure, it can only be qualitative due each procedure being different. Variables for each procedure include (but not limited) the following: Clinical condition of patient, product type used, point of entry site, skill of user.